CLINICAL TRIAL: NCT03132701
Title: The Effect of Magnesium Supplementation During General Anesthesia on the Quality of Postoperative Recovery in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H1703-110-840
Record Dates: First submitted 2017-04-09; First posted 2017-04-28 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Emergence Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Magnesium; Magnesium Sulfate; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium group (Active Comparator): Mg is administered with dose of 30 mg/kg for 10 minutes and then 10 mg/kg/hr until 5 minutes before surgery ends
  Interventions: Drug: Magnesium
- Control group (Placebo Comparator): Saline is administered with same volume of Mg of magnesium group until 5 minutes before surgery ends
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Magnesium — Mg is administered during anesthesia until 5 minutes before surgery ends
  Other Names: Magnesium sulfate
  Arms: Magnesium group
Drug: Saline — Same volume of saline is infused until 5 minutes before surgery ends
  Other Names: Normal saline
  Arms: Control group

SUMMARY:
Evaluation of prevention of emergence delirium and analgesic effect of magnesium on children

DETAILED DESCRIPTION:
Children < 8 years old who scheduled for elective opthalmic surgery are randomly assigned to Magnesium (Mg) group and control group. Before anesthetic induction, modified Yale Preoperative Anxiety Scale (m-YPAS) is assessed. Routine anesthetic induction is performed, and neuromuscular blocker is not used. Laryngeal mask airway is inserted and controlled ventilation is started.

In Mg group, Mg of 30 mg/kg is administered for 10 minutes and then continuously infused (10mg/kg/hr) until 5 minutes before surgery end. In control group, the similar volume of saline is infused.

Pediatric Anesthesia Emergence Delirium (PAED) scale and pain score (Modified Children's Hospital of Eastern Ontario Pain Scale, CHEOPS) will be measured immediately after and 30 minutes after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 2 and 7 years
* American Society of Anesthesiologist physical status 1 and 2
* Children scheduled for opthalmic surgery

Exclusion Criteria:

* Allergy history to any drugs
* Risk of malignant hyperthermia
* Neuromuscular disease
* With arrhythmia
* Any pulmonary, cardiac, hepatic and renal disease
* Obesity

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Emergence delirium | 30 minutes after anesthesia
  Pediatric Anesthesia Emergence Delirium (PAED) scale

SECONDARY OUTCOMES:
Pain score | At each two points: during emergence in operating room and 30 minutes after surgery ends
  Modified Children's Hospital of Eastern Ontario Pain Scale, CHEOPS)
Nausea | At each two points: during emergence in operating room and 30 minutes after surgery ends
  visual analogue scale
vomiting | At each two points: during emergence in operating room and 30 minutes after surgery ends
  number
Duration of post-anesthetic care unit (PACU) stay | During 1 hour after surgery at PACU
  Duration of post-anesthetic care unit (PACU) stay

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- SNUH, Seoul, Jongro Gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee JH, Choi S, Lee M, Jang YE, Kim EH, Kim JT, Kim HS. Effect of magnesium supplementation on emergence delirium and postoperative pain in children undergoing strabismus surgery: a prospective randomised controlled study. BMC Anesthesiol. 2020 Nov 18;20(1):289. doi: 10.1186/s12871-020-01192-7. PMID 33208099